CLINICAL TRIAL: NCT01070914
Title: The Israeli National Consortium for Early Detection and Characterization of Primary Ciliary Dyskinesia
Brief Title: Early Detection and Characterization of Primary Ciliary Dyskinesia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Collaborators: Rambam Health Care Campus (Other); Hadassah Medical Organization (Other); Tel-Aviv Sourasky Medical Center (Other Government); Sheba Medical Center (Other Government); Assaf-Harofeh Medical Center (Other Government); The Nazareth Hospital, Israel (Other); Soroka University Medical Center (Other); Shaare Zedek Medical Center (Other); Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: Hackmon-2
Record Dates: First submitted 2010-02-06; First posted 2010-02-18 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: Cilia; Phenotyping; Diagnosis; Nitric Oxide; Bronchiectasis
MeSH Terms: conditions — Ciliary Motility Disorders; Disease; Bronchiectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Primary Ciliary Dyskinesia (PCD) is a severe genetic disorder caused by various mutations in genes affecting ciliary motility. Various new and complementary diagnostic techniques, including measurements of nasal nitric oxide (NO), Video Microscopy (VM), Immunoflourescence (IF) and genetic analysis have recently been recognized as simpler and more accurate modalities for the diagnosis and characterization of patients with PCD compared to electron microscopy. While considered a rare disease worldwide, PCD is more prevalent among highly consanguineous populations, such as those found in Israel. We hypothesize that using modern state of the art and novel test modalities on a national scale in Israel will improve diagnosis, improve phenotypic-genotypic correlations and create a national registry for PCD.

DETAILED DESCRIPTION:
Primary Ciliary Dyskinesia (PCD) is a severe genetic disorder caused by various mutations in genes affecting ciliary motility. While diagnosis of PCD in Israel is currently based for the most part on electron microscopy (EM) detection of ciliary ultrastructural defects, this technique may be unsatisfactory and does not overcome the inherent heterogeneity. Thus, late and under-diagnosis and suboptimal characterization of patients is common. Various newer and complementary diagnostic techniques, including measurements of nasal nitric oxide (NO), Video Microscopy (VM), Immunoflourescence (IF) and genetic analysis have recently been recognized as simpler and more accurate modalities for the diagnosis and characterization of patients with PCD. While considered a rare disease worldwide, PCD is more prevalent among highly consanguineous populations, such as those found in Israel. Given the rarity of cases particularly familial ones, the most useful implementation of new diagnostic techniques requires multicenter collaboration.

We hypothesize that using modern state of the art and novel test modalities on a national scale in Israel will improve diagnosis, improve phenotypic-genotypic correlations and create a national registry for PCD.

We propose to perform such a multicenter study whose aims are:

* To characterize the complex phenotype and genotype of PCD in Israel, using state-of-the-art and novel diagnostic techniques.
* To create a national registry of patients and families with PCD in Israel
* To develop robust national standards of diagnosis and evaluation, which will lead to better and earlier diagnosis, treatment and counseling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCD diagnosis
* Subjects with suspected diagnosis of PCD

Exclusion Criteria:

* Subjects Uncooperative with study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents of Israel
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Phenotypic and genetic characterization | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — Ziv Medical Center
Locations (1):
- Ziv Medical center, Safed, Israel

REFERENCES:
- [Derived] Amirav I, Mussaffi H, Roth Y, Schmidts M, Omran H, Werner C; Israeli PCD Consortium Investigators. A reach-out system for video microscopy analysis of ciliary motions aiding PCD diagnosis. BMC Res Notes. 2015 Mar 8;8:71. doi: 10.1186/s13104-015-0999-x. PMID 25869032